CLINICAL TRIAL: NCT02753920
Title: A Randomized, Controlled Trial After Vaginal Apex Suspension Comparing Force of Stream to Traditional Retrograde Fill Voiding Trial
Brief Title: Comparing Force of Stream to Retrograde Fill Voiding Trial After Vaginal Apex Suspension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, Harvey Winkler, Co-Chief, Northwell Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HS16-0232
Record Dates: First submitted 2016-04-12; First posted 2016-04-28 (Estimated); Results first posted 2018-11-05 (Actual); Last update posted 2018-11-05 (Actual); Status verified 2018-11

CONDITIONS: Vaginal Apical Prolapse
Keywords: voiding trial; prolapse
MeSH Terms: conditions — Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Retrograde fill voiding trial method (Active Comparator): 1. Bladder drained with indwelling foley catheter, then retrograde filled with 300cc sterile water.
  2. Catheter is removed
  3. Patient voids within 20 minutes (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction).
  4. The patient will subjectively quantify their force of stream via visual analog scale (VAS) scale (however this information will only be used for research purposes).
  5. If she voids >/= 2/3 (200cc) the catheter will remain out as she will have passed her voiding trial. If she voids <200cc she will be discharged home with a catheter and instructed to follow-up in 2-5 days for an in-office retrograde voiding trial.
  Interventions: Other: voiding trial; Device: Foley catheter
- Force of Stream (FAST) voiding trial method (Active Comparator): 1. Bladder drained with indwelling foley catheter, then retrograde filled with 300cc sterile water.
  2. Catheter is removed
  3. Patient voids within 20 minutes (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction).
  4. The patient will subjectively quantify their force of stream via VAS scale.
  5. If VAS scale >/=50 (>/=50%) the catheter will remain out, patient is discharged home without measuring a PVR
  6. If VAS scale is from 0-49 (=0-49%) a PVR will be checked via bladder scan. If PVR is <500cc, the patient will be discharged without a catheter; if PVR is >/=500cc, the patient will be discharged with a catheter. If she is discharged with an indwelling foley catheter, she will have an in-office retrograde voiding trial in 2-5 days.
  Interventions: Other: voiding trial; Device: Foley catheter

INTERVENTIONS:
Other: voiding trial — 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling
Device: Foley catheter — If subject is unable to void adequately, a Foley catheter will be placed as per protocol and the subject discharged home with catheter. The subject will follow up in the office for removal of catheter.

SUMMARY:
Voiding difficulties are common after prolapse and incontinence surgeries. All patients after vaginal prolapse surgery must complete a voiding trial if they are to be discharged home without a catheter. Accepted protocols for voiding trials after prolapse and incontinence surgeries do not exist. The purpose of this study is to compare two different types of postoperative voiding trials to determine which leads to less postoperative issues, such as urinary retention requiring catheterization. You are being asked to participate because you are having a vaginal apex suspension surgery.

DETAILED DESCRIPTION:
It is common to have voiding difficulties after prolapse and incontinence surgeries. Difficulties in voiding are seen in up to 47% of patients after transvaginal prolapse surgery in the immediate hours postoperatively (6). Accepted protocols for voiding trials after prolapse and incontinence surgeries do not exist. Traditionally, many surgeons measure postvoid residual (PVR) urine volume to assess incomplete bladder emptying by retrograde filling the bladder with a predetermined amount of normal saline or water. The catheter is then removed and the patient is permitted to void into a collection basin. The need for postoperative catheterization is generally based on arbitrarily determined ratios of voided urine to PVR. The force of stream trial (FAST) does not prioritize amount voided, but rather the patient's subjective force of stream. Using FAST, a patient uses a visual analog scale (VAS) scale to quantify her force of stream. If she states that her Force of Stream (FOS) is >50% of her baseline prior to surgery, independent of the amount voided, she is discharged without a catheter. If the FOS is <50%, a PVR is measured via bladder scan. If her PVR is <500cc the patient is discharged home.

No randomized control trials (RCT) have been performed comparing the FAST method to the traditional retrograde voiding trial in subjects undergoing vaginal apex prolapse surgery despite the promising findings that FAST voiding trials are as reliable and safe as retrograde voiding trials in patients undergoing anti-incontinence surgeries. Standard in our practice is to perform a voiding trial on postoperative day 1 on all patients after vaginal apical prolapse surgery if they are to be discharged without a catheter. Investigators would like to compare the FAST voiding trial to a traditional retrograde fill voiding trial with respect to the rate of catheterization among those discharged without a catheter within the six-week postoperative period in patients undergoing a vaginal apex prolapse surgery. Investigators hypothesize the FAST voiding trial method is not inferior to traditional retrograde voiding trial. Subjects will complete questionnaires to examine postoperative bladder function, symptom distress and quality of life before and after surgery during their routine postoperative visits.

ELIGIBILITY:
Inclusion Criteria:

1. Women undergoing vaginal apex surgery (sacrocolpopexy, sacrospinous ligament suspension, uterosacral ligament suspension, colpocleisis) with or without mid-urethral sling, with or without anterior or posterior colporrhaphy

Exclusion Criteria:

1. Patients who underwent a surgery that requires long term catheterization (i.e fistula repair or urethral diverticulum)
2. Patients who sustained a cystotomy during surgery as our divisional protocol is to send these patients home with a Foley catheter for 5-14 days without a voiding trial
3. Patients with baseline urinary retention and the inability to urinate without catheterization
4. Pregnant women

Ages: 18 Years to 95 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 184 (Actual)
Dates: Start 2016-03; Primary Completion 2017-06 (Actual); Study Completion 2018-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Northwell Health System Division of Urogynecology, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Swift S, Woodman P, O'Boyle A, Kahn M, Valley M, Bland D, Wang W, Schaffer J. Pelvic Organ Support Study (POSST): the distribution, clinical definition, and epidemiologic condition of pelvic organ support defects. Am J Obstet Gynecol. 2005 Mar;192(3):795-806. doi: 10.1016/j.ajog.2004.10.602. PMID 15746674
- [Background] Swift SE. The distribution of pelvic organ support in a population of female subjects seen for routine gynecologic health care. Am J Obstet Gynecol. 2000 Aug;183(2):277-85. doi: 10.1067/mob.2000.107583. PMID 10942459
- [Background] Smith FJ, Holman CD, Moorin RE, Tsokos N. Lifetime risk of undergoing surgery for pelvic organ prolapse. Obstet Gynecol. 2010 Nov;116(5):1096-100. doi: 10.1097/AOG.0b013e3181f73729. PMID 20966694
- [Background] Stav K, Dwyer PL, Rosamilia A, Schierlitz L, Lim YN, Chao F, De Souza A, Thomas E, Murray C, Conway C, Lee J. Repeat synthetic mid urethral sling procedure for women with recurrent stress urinary incontinence. J Urol. 2010 Jan;183(1):241-6. doi: 10.1016/j.juro.2009.08.111. PMID 19913831
- [Background] Turner LC, Kantartzis K, Shepherd JP. Predictors of postoperative acute urinary retention in women undergoing minimally invasive sacral colpopexy. Female Pelvic Med Reconstr Surg. 2015 Jan-Feb;21(1):39-42. doi: 10.1097/SPV.0000000000000110. PMID 25185611
- [Background] Foster RT Sr, Borawski KM, South MM, Weidner AC, Webster GD, Amundsen CL. A randomized, controlled trial evaluating 2 techniques of postoperative bladder testing after transvaginal surgery. Am J Obstet Gynecol. 2007 Dec;197(6):627.e1-4. doi: 10.1016/j.ajog.2007.08.017. PMID 18060956
- [Background] Kleeman S, Goldwasser S, Vassallo B, Karram M. Predicting postoperative voiding efficiency after operation for incontinence and prolapse. Am J Obstet Gynecol. 2002 Jul;187(1):49-52. doi: 10.1067/mob.2002.124841. PMID 12114887
- [Background] Pulvino JQ, Duecy EE, Buchsbaum GM, Flynn MK. Comparison of 2 techniques to predict voiding efficiency after inpatient urogynecologic surgery. J Urol. 2010 Oct;184(4):1408-12. doi: 10.1016/j.juro.2010.05.096. Epub 2010 Aug 19. PMID 20727543
- [Background] Ingber MS, Vasavada SP, Moore CK, Rackley RR, Firoozi F, Goldman HB. Force of stream after sling therapy: safety and efficacy of rapid discharge care pathway based on subjective patient report. J Urol. 2011 Mar;185(3):993-7. doi: 10.1016/j.juro.2010.10.050. Epub 2011 Jan 19. PMID 21247598
- [Background] Tunitsky-Bitton E, Murphy A, Barber MD, Goldman HB, Vasavada S, Jelovsek JE. Assessment of voiding after sling: a randomized trial of 2 methods of postoperative catheter management after midurethral sling surgery for stress urinary incontinence in women. Am J Obstet Gynecol. 2015 May;212(5):597.e1-9. doi: 10.1016/j.ajog.2014.11.033. Epub 2014 Nov 27. PMID 25434837
- [Background] Peleg AY, Hooper DC. Hospital-acquired infections due to gram-negative bacteria. N Engl J Med. 2010 May 13;362(19):1804-13. doi: 10.1056/NEJMra0904124. No abstract available. PMID 20463340
- [Background] Elkadry EA, Kenton KS, FitzGerald MP, Shott S, Brubaker L. Patient-selected goals: a new perspective on surgical outcome. Am J Obstet Gynecol. 2003 Dec;189(6):1551-7; discussion 1557-8. doi: 10.1016/s0002-9378(03)00932-3. PMID 14710061
- [Background] Sutkin G, Lowder JL, Smith KJ. Prophylactic antibiotics to prevent urinary tract infection during clean intermittent self-catheterization (CISC) for management of voiding dysfunction after prolapse and incontinence surgery: a decision analysis. Int Urogynecol J Pelvic Floor Dysfunct. 2009 Aug;20(8):933-8. doi: 10.1007/s00192-009-0885-y. Epub 2009 Apr 10. PMID 19582384
- [Background] Chung CP, Kuehl TJ, Harris SK, McBride MM, Larsen WI, Yandell PM, Shull BL. Incidence and risk factors of postoperative urinary tract infection after uterosacral ligament suspension. Int Urogynecol J. 2012 Jul;23(7):947-50. doi: 10.1007/s00192-012-1709-z. Epub 2012 Mar 8. PMID 22398827
- [Background] Barber MD, Kleeman S, Karram MM, Paraiso MF, Walters MD, Vasavada S, Ellerkmann M. Transobturator tape compared with tension-free vaginal tape for the treatment of stress urinary incontinence: a randomized controlled trial. Obstet Gynecol. 2008 Mar;111(3):611-21. doi: 10.1097/AOG.0b013e318162f22e. PMID 18310363
- [Background] Ward KL, Hilton P; UK and Ireland TVT Trial Group. Tension-free vaginal tape versus colposuspension for primary urodynamic stress incontinence: 5-year follow up. BJOG. 2008 Jan;115(2):226-33. doi: 10.1111/j.1471-0528.2007.01548.x. Epub 2007 Oct 25. PMID 17970791
- [Background] Liapis A, Bakas P, Creatsas G. Long-term efficacy of tension-free vaginal tape in the management of stress urinary incontinence in women: efficacy at 5- and 7-year follow-up. Int Urogynecol J Pelvic Floor Dysfunct. 2008 Nov;19(11):1509-12. doi: 10.1007/s00192-008-0664-1. Epub 2008 Jun 10. PMID 18542836
- [Derived] Pilkinton ML, Williams KS, Sison CP, Shalom DF, Winkler HA. Comparing Force of Stream With a Standard Fill Voiding Trial After Surgical Repair of Apical Prolapse: A Randomized Controlled Trial. Obstet Gynecol. 2019 Apr;133(4):675-682. doi: 10.1097/AOG.0000000000003159. PMID 30870290

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After signing informed consent and enrolling in the study, 4 subjects withdrew consent prior to randomization, 4 subjects had surgery cancelled for various medical reasons, 3 subjects had cystotomies thus requiring prolonged catheterization for 1-2 weeks and 1 subject withdrew after randomization.
Groups:
- Retrograde Fill Voiding Trial Method: Bladder drained w/ indwelling foley catheter, then retrograde filled w/ 300cc sterile water. Catheter is removed. Patient voids w/in 20 min (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction). Patient subjectively quantify their force of stream via visual analog scale (VAS) scale (however this information will only be used for research purposes). If she voids >/= 2/3 (200cc) the catheter will remain out as she will have passed her voiding trial. If she voids <200cc she will be discharged home with a catheter and instructed to follow-up in 2-5 days for an in-office retrograde voiding trial.
  TOV (trial of void): 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling. catheter: If subject unable to void adequately, a Foley catheter will be placed as per protocol and the subject discharged home with catheter.
- Force of Stream (FAST) Voiding Trial Method: Bladder drained w/ indwelling foley catheter, then retrograde filled w/ 300cc sterile water. Catheter is removed. Patient voids w/in 20 minutes (if unable to void after 20 minutes, discharged home w/ a catheter secondary to voiding dysfunction). The patient will subjectively quantify their force of stream via VAS scale. If VAS scale >/=50 (>/=50%) the catheter will remain out, patient is discharged home without measuring a PVR (postvoid residual). If VAS scale is from 0-49 (=0-49%) a PVR will be checked via bladder scan. If PVR is <500cc, the patient will be discharged without a catheter; if PVR is >/=500cc, the patient will be discharged with a catheter. If she is discharged with an indwelling foley catheter, she will have an in-office retrograde voiding trial in 2-5 days TOV: 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling catheter: If subject is unable to void adequately
Period: Overall Study
Arm/Group | Retrograde Fill Voiding Trial Method | Force of Stream (FAST) Voiding Trial Method
Started | 87 | 86
Completed | 87 | 86
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Retrograde Fill Voiding Trial Method: Bladder drained w/indwelling foley catheter, then retrograde filled with 300cc sterile water. Catheter removed. \Patient voids within 20 minutes (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction). Patient subjectively quantify their force of stream via visual analog scale (VAS) scale (however this information will only be used for research purposes). If she voids >/= 2/3 (200cc) catheter will remain out as she will have passed her voiding trial. If she voids <200cc she will be discharged home with a catheter and instructed to follow-up in 2-5 days for an in-office retrograde voiding trial.
  TOV: 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling Foley catheter: If subject is unable to void adequately, a Foley catheter will be placed as per protocol and the subject discharged home with catheter. Subject will follow up in the office for removal of catheter.
- Force of Stream (FAST) Voiding Trial Method: Bladder drained with foley catheter, then retrograde filled with 300cc sterile water. Catheter removed. Patient voids within 20 min (if unable to void after 20 min, she discharged home w/catheter secondary to voiding dysfunction). Patient subjectively quantify their force of stream via VAS scale. If VAS scale >/=50 (>/=50%) catheter will remain out, patient is discharged home w/o measuring a PVR If VAS scale is from 0-49 (=0-49%) PVR checked via bladder scan. If PVR is <500cc, patient discharged w/o catheter; if PVR is >/=500cc, patient discharged w/catheter. If discharged with an indwelling foley catheter, she will have an in-office retrograde voiding trial in 2-5 days.
  TOV: 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling Foley catheter: If subject unable to void adequately, Foley catheter placed as per protocol and subject discharged home with catheter. Subject follow up in the office for removal of catheter.
- Total: Total of all reporting groups
Arm/Group | Retrograde Fill Voiding Trial Method | Force of Stream (FAST) Voiding Trial Method | Total
Number analyzed (Participants) | 87 | 86 | 173
Age, Continuous [Median (Standard Deviation); unit: years] | 63.1 (11.4) | 62.7 (10.5) | 62.9 (11.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  female | 87 | 86 | 173
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 8 | 18
  Not Hispanic or Latino | 77 | 78 | 155
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects Catheterized Within the Six-week Post-operative Period Following Surgical Repair of Prolapse, Among Those Discharged Without a Urinary Catheter.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Retrograde Fill Voiding Trial Method | Force of Stream (FAST) Voiding Trial Method
Number analyzed (Participants) | 64 | 71
Participants | 2 | 2

2. Secondary Outcome: Number of Subjects Discharged With a Catheter (This is Essentially the Proportion of Patients Who Failed the Voiding Trial)
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Groups:
- Retrograde Fill Voiding Trial Method: Bladder drained w/ indwelling foley catheter, then retrograde filled w/ 300cc sterile water. Catheter is removed. Patient voids w/in 20 min (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction). Patient subjectively quantify their force of stream via visual analog scale (VAS) scale (however this information will only be used for research purposes). If she voids >/= 2/3 (200cc) the catheter will remain out as she will have passed her voiding trial. If she voids <200cc she will be discharged home with a catheter and instructed to follow-up in 2-5 days for an in-office retrograde voiding trial.
  TOV: 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling. catheter: If subject unable to void adequately, a Foley catheter will be placed as per protocol and the subject discharged home with catheter.
- Force of Stream (FAST) Voiding Trial Method: Bladder drained w/ indwelling foley catheter, then retrograde filled w/ 300cc sterile water. Catheter is removed. Patient voids w/in 20 minutes (if unable to void after 20 minutes, discharged home w/ a catheter secondary to voiding dysfunction). The patient will subjectively quantify their force of stream via VAS scale. If VAS scale >/=50 (>/=50%) the catheter will remain out, patient is discharged home without measuring a PVR. If VAS scale is from 0-49 (=0-49%) a PVR will be checked via bladder scan. If PVR is <500cc, the patient will be discharged without a catheter; if PVR is >/=500cc, the patient will be discharged with a catheter. If she is discharged with an indwelling foley catheter, she will have an in-office retrograde voiding trial in 2-5 days TOV: 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling catheter: If subject is unable to void adequately
Arm/Group | Retrograde Fill Voiding Trial Method | Force of Stream (FAST) Voiding Trial Method
Number analyzed (Participants) | 87 | 86
Participants | 23 | 15

3. Secondary Outcome: Proportion of Patients With Unexpected Visits to the Clinic, Within the Six-week Post-operative Period.
Time Frame: 6 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Force of Stream (FAST) Voiding Trial Method | Retrograde Fill Voiding Trial Method
Number analyzed (Participants) | 86 | 87
Participants | 8 | 6

ADVERSE EVENTS:
Time Frame: 6 weeks postoperatively.
Groups:
- Retrograde Fill Voiding Trial Method: Bladder drained with indwelling foley catheter, then retrograde filled with 300cc sterile water. Catheter is removed Patient voids w/in 20 minutes (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction). patient subjectively quantify their force of stream via visual analog scale (VAS) scale (however information will only be used for research purposes).
  If she voids >/= 2/3 (200cc) catheter will remain out as she will have passed her voiding trial. If she voids <200cc she will be discharged home with a catheter and instructed to follow-up in 2-5 days for an in-office retrograde voiding trial.
  TOV: 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling catheter: If subject is unable to void adequately, a Foley catheter will be placed as per protocol and the subject discharged home with catheter. The sub
- Force of Stream (FAST) Voiding Trial Method: Bladder drained with indwelling foley catheter, then retrograde filled with 300cc sterile water. Catheter is removed Patient voids within 20 minutes (if unable to void after 20 minutes, she will be discharged home with a catheter secondary to voiding dysfunction). The patient will subjectively quantify their force of stream via VAS scale. If VAS scale >/=50 (>/=50%) catheter will remain out, patient discharged home without measuring a PVR. If VAS scale is from 0-49 (=0-49%) a PVR will be checked via bladder scan. If PVR is <500cc, the patient will be discharged without a catheter; if PVR is >/=500cc, patient discharged with a catheter. If she is discharged with an indwelling foley catheter, she will have an in-office retrograde voiding trial in 2-5 days.
  voiding trial: 1 of 2 tests to assess bladder function after vaginal apex suspension surgery with or without mid-urethral sling
  Foley catheter: If subject is unable to void adequately
Arm/Group | Retrograde Fill Voiding Trial Method | Force of Stream (FAST) Voiding Trial Method
All-Cause Mortality (participants affected / at risk) | 0/87 | 0/86
Serious Adverse Events (participants affected / at risk) | 0/87 | 0/86
Other Adverse Events (participants affected / at risk) | 0/87 | 0/86

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-02-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT02753920/Prot_SAP_000.pdf